CLINICAL TRIAL: NCT00995657
Title: Dose Response of FENO to Inhaled Steroids in Mild-to-moderate Asthma
Brief Title: Dose Response of Fractional Exhaled Nitric Oxide (FeNO) to Inhaled Steroids in Mild-to-moderate Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PAW003
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose ICS (Active Comparator): Fluticasone Propionate 250mcg bid
  Interventions: Drug: Fluticasone Propionate
- Low dose ICS (Active Comparator): Fluticasone propionate 50mcg bid
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate — Inhaled Fluticasone Propionate 50mcg bid
  Arms: Low dose ICS
Drug: Fluticasone Propionate — Inhaled Fluticasone Propionate 250mcg bid
  Arms: High dose ICS

SUMMARY:
Asthma is a chronic disease, which means that it cannot be cured, but the investigators can use inhalers and tablets to control the symptoms. In asthma, the airways become inflamed and irritated which can cause coughing and make the airways tighten. This 'inflammation' is the root of the problem in asthma. Doctors have different ways to measure the inflammation in the airways. One way is to measure a gas called nitric oxide (NO) on the breath. This is made by the lungs when asthmatic inflammation is present. The investigators have been using NO as a test in research labs for many years, but there are still unanswered questions about how it changes between morning and night and how quickly medicines work on it. In most asthmatics, even small doses of inhaled steroids (preventers) can reduce the NO levels to normal, but in some people this does not seem to happen. The investigators now have portable NO machines that are designed for patients to use in the home. The investigators want to follow NO readings in patients with high levels to measure how they respond to different doses of steroid inhalers. The investigators hope this will help the investigators better understand asthma inflammation and treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis os asthma, taking 200-1000mcg budesonide or equivalent per day
* FENO greater than 30ppb on treatment

Exclusion Criteria:

* Recent RTI or prednisolone
* Smoking within 1 year or 10 pack years
* ABPA, COPD, bronchiectasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in FENO | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Williamson, MBChB, Principal Investigator — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, University of Dundee, Dundee, Tayside, United Kingdom

REFERENCES:
- [Result] Anderson WJ, Short PM, Williamson PA, Lipworth BJ. Inhaled corticosteroid dose response using domiciliary exhaled nitric oxide in persistent asthma: the FENOtype trial. Chest. 2012 Dec;142(6):1553-1561. doi: 10.1378/chest.12-1310. PMID 23364390
- [Derived] Anderson WJ, Short PM, Jabbal S, Lipworth BJ. Inhaled corticosteroid dose response in asthma: Should we measure inflammation? Ann Allergy Asthma Immunol. 2017 Feb;118(2):179-185. doi: 10.1016/j.anai.2016.11.018. Epub 2017 Jan 3. PMID 28065396